CLINICAL TRIAL: NCT04714190
Title: Randomized, Controlled, Multicenter Phase III Clinical Study Evaluating the Efficacy and Safety of RC48-ADC for the Treatment of Locally Advanced or Metastatic Gastric Cancer With HER2-overexpression
Brief Title: A Study of RC48-ADC in Local Advanced or Metastatic Gastric Cancer With the HER2-Overexpression
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C007
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Gastric Cancer; HER2 Overexpressing Gastric Carcinoma
Keywords: RC48-ADC; HER2 overexpression; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Injections; Paclitaxel; Irinotecan; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RC48-ADC (Experimental): Participants will receive RC48-ADC every 2 weeks (Q2W) until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: RC48-ADC
- Physician's Choice (Active Comparator): Participants will receive physician choosed chemotherapy from the following options: Paclitaxel Injection or Irinotecan Hydrochloride Injection or Apatinib Mesylate Tablets oral.
  Interventions: Drug: Paclitaxel injection; Drug: Irinotecan Hydrochloride Injection; Drug: Apatinib Mesylate Tablets

INTERVENTIONS:
Drug: RC48-ADC — 2.5 mg/kg IV every 2 weeks
  Other Names: Recombinant Humanized anti-HER2 Monoclonal Antibody-MMAE Conjugate For Injection
  Arms: RC48-ADC
Drug: Paclitaxel injection — Administered according to label, as one option for Physician's Choice (determined before randomization)
  Other Names: Taxol
  Arms: Physician's Choice
Drug: Irinotecan Hydrochloride Injection — Administered according to label, as one option for Physician's Choice (determined before randomization)
  Other Names: CAMPTO
  Arms: Physician's Choice
Drug: Apatinib Mesylate Tablets — Administered according to label, as one option for Physician's Choice (determined before randomization)
  Other Names: Aitan
  Arms: Physician's Choice

SUMMARY:
This is a Phase III, randomized, multicenter, open-label clinical trial designed to compare RC48-ADC to physician choice standard treatment in participants with human epidermal growth factor receptor 2 (HER2)-overexpression locally advanced or metastatic gastric cancer.

DETAILED DESCRIPTION:
This study is a phase III multi-center, randomized, open-label, parallel control study to evaluate the efficacy and safety of recombinant humanized anti-HER2 monoclonal antibody-Monomethyl auristatin E (MMAE) conjugate for the treatment of HER2-overexpression locally advanced or metastatic gastric cancer. The HER2-overexpression is defined as: the HER2 IHC 3+ or 2+, regardless of FISH status.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Male or female, Age ≥ 18 years.
* Predicted survival ≥ 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* All female subjects will be considered to be of child-bearing potential unless they are postmenopausal, or have been sterilized surgically.Female subjects of child-bearing potential must agree to use two forms of highly effective contraception. Male subjects and their female partner who are of child-bearing potential must agree to use two forms of highly effective contraception.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.
* Adequate organ function.
* All subjects must have inoperable, advanced or metastatic gastric or or gastroesophageal adenocarcinoma
* Have had progression or intolerance following receipt of at least two systemic chemotherapy for advanced or metastatic disease.
* The HER2 IHC test result is IHC 2+ or IHC 3+, the subject's previous test results (confirmed by the investigator) or the research center's test results are acceptable; the subject can provide the Specimen of primary or metastatic tumor for HER2 review/judgment.
* HER2 classic positive (definition: IHC3+ or IHC2+FISH+) and patients who have previously failed standard treatment
* According to the RECIST 1.1 standard, there is at least one measurable lesion.

Exclusion Criteria:

* Known hypersensitivity to Recombinant Humanized Anti-HER2 Monoclonal Antibody-MMAE Conjugate For Injection.
* History of receiving any anti-cancer drug/biologic treatment within 4 weeks prior to trial treatment.
* History of major surgery within 4 weeks of planned start of trial treatment.
* Has received a live virus vaccine within 4 weeks of planned start of trial treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or cancers with a similar curative outcome as those mentioned above.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | within approximately 3 years
  Overall survival (OS) refers to the time from the date of randomization to the date of death of the subject.

SECONDARY OUTCOMES:
Progression-free survival (PFS), evaluated by the investigator | within approximately 3 years
  Progression-free survival (PFS) refers to the time from the date of randomization to the first researcher's evaluation of disease progression or death (calculated by the event that occurred first). The disease progression will be evaluated by the researchers according to the RECIST 1.1 standard.
Objective remission rate (ORR) | within approximately 3 years
  The objective response rate will be mainly analyzed by the independent efficacy evaluation committee according to the RECIST 1.1 standard tumor evaluation (the evaluation by the investigator will also be performed).
Duration of relief (DOR) | within approximately 3 years
  DOR is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death
Disease control rate (DCR) | within approximately 3 years
  Disease control rate (DCR) is defined as cases where objective remission (assessed as complete remission or partial remission according to RECIST 1.1 standard) or stable disease during the study.
Tumor progression time (TTP) | within approximately 3 years
  Time to disease progression (TTP) refers to the time from the random date to the first disease progression (calculated by the event that occurred first). Disease progression will be evaluated by the investigator according to the RECIST 1.1 standard (investigator and Independent Review Committee(IRC) evaluation).

CONTACTS AND LOCATIONS:
Locations (52):
- China (52):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Affiliated Hospital of Hebei University, Baoding
  - China-Japan Friendship Hospital, Beijing
  - Luhe Hospital Affiliated to Capital Medical University, Beijing
  - Peking University People's Hospital, Beijing
  - Jilin Provincial Tumor Hospital, Changchun
  - Xiangya Hospital of Central South University, Changsha
  - Affiliated Hospital of Chengde Medical College, Chengde
  - Three Gorges Hospital Affiliated to Chongqing University, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Southern Hospital of Southern Medical University, Guangzhou
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - The Affiliated Tumor Hospital of Harbin Medical University, Harbin
  - Anhui Cancer Hospital, Hefei
  - Anhui Provincial Hospital, Hefei
  - Jinan Central Hospital, Jinan
  - Shandong Cancer Hospital, Jinan
  - Affiliated Hospital of Jining Medical College, Jining
  - The First People's Hospital of Jining City, Jining
  - Lanzhou University Second Hospital, Lanzhou
  - Linyi Tumor Hospital, Linyi
  - Drum Tower Hospital Affiliated to Nanjing University School of Medicine, Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - The First Affiliated Hospital of Nanjing Medical University (Jiangsu Provincial People's Hospital), Nanjing
  - Qingdao University Hospital, Qingdao
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Changhai Hospital, Shanghai
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai
  - Cancer Hospital Affiliated to Shantou University Medical College, Shantou
  - Liaoning Cancer Hospital, Shenyang
  - Shenzhen People's Hospital, Shenzhen
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Shanxi Cancer Hospital, Taiyuan
  - Tianjin Cancer Hospital, Tianjin
  - Weifang People's Hospital, Weifang
  - Weihai Municipal Hospital, Weihai
  - Huazhong University of Science Tongji Hospital, Tongji Medical College, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Affiliated Hospital of Qinghai University, Xining
  - Qinghai Provincial People's Hospital, Xining
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Xuzhou Central Hospital, Xuzhou
  - Subei People's Hospital of Jiangsu Province, Yangzhou
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou